CLINICAL TRIAL: NCT07301541
Title: Test, Validation and Implementation of a Screening Tool (STOB) for the Early Detection of Binge Eating Disorder (BED) and Insights Into BE Development in Children and Adolescents Participating in a Multicomponent Camp Intervention With or Without a Parental BED Intervention
Brief Title: Screening for Binge Eating Disorder and Insights Into BE Behavior in Children and Adolescents Participating in a Multicomponent Camp Intervention With or Without a Parental BED Intervention
Acronym: STOB
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Julemærkefonden (Unknown); Danish National Center for Obesity, Aarhus University Hospital, Denmark (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STOB 2.0; Journal number 05-0801-2595 (Other Grant/Funding Number: The Danish Health Authority)
Record Dates: First submitted 2025-11-28; First posted 2025-12-24 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-11

CONDITIONS: Binge Eating Disorder; Binge Eating; Loss of Control Eating; Overweight , Obesity; Children; Childhood Obesity; Screening; BED
Keywords: Binge eating; Binge eating disorder; Lifestyle intervention; Children; Loss of control eating; Adolescents; BED; Screening
MeSH Terms: conditions — Binge-Eating Disorder; Bulimia; Overweight; Obesity; Pediatric Obesity

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Masking Description: Camp staff have no knowledge of or influence on which parents/guardians are assigned to the parent-based BED intervention. Study staff performing the ChEDE after the camp intervention will be blinded to group assignment.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard parent involvement during camp (P-ST) (Active Comparator): Parents or guardians will receive the standard parental involvement during and in relation to their child's camp attendance. This includes individual meetings with camp staff and parental educational days focused on gaining insight into camp life, as well as participating in social and physical activities and cooking classes.
  Interventions: Behavioral: A 10-week multicomponent camp intervention for children
- Add-on parent-based BED intervention during camp (P-BED) (Experimental): In addition to the standard parental involvement (P-ST) during camp, parents/guardians will receive a virtual parent-based BED intervention during the 10-week their child attend camp. The intervention will be designed to provide knowledge about BED and tools to support their child's eating after the intervention.
  Interventions: Behavioral: A 10-week multicomponent camp intervention for children; Behavioral: A BED intervention for parents

INTERVENTIONS:
Behavioral: A 10-week multicomponent camp intervention for children — A 10-week multicomponent camp intervention for participating children only, focusing on social and physical activities, healthy meals, and daily physical activities.
Behavioral: A BED intervention for parents — An add-on virtual parent-based intervention providing knowledge about BED and tools to support their child's eating after the multicomponent camp intervention.
  Arms: Add-on parent-based BED intervention during camp (P-BED)

SUMMARY:
The main purpose is to investigate the effectiveness of a 10-week multicomponent camp intervention to reduce BE behavior in children and adolescents and explore in a randomized controlled setting if a parent-based BED-intervention has any add-on effect, attenuating the development of BE behavior in this sample. The study will include an initial follow-up assessment scheduled 10-12 weeks after camp completion and plans for long-term follow-up assessments two and five years after inclusion.

Overall, we hypothesize that the multicomponent camp intervention will effectively reduce BE behavior in children and adolescents. Furthermore, we hypothesize that participants whose parents are randomized to receive the parental BED intervention will show a lower prevalence of BE behavior one year after the camp intervention compared with children whose parents receive standard care.

DETAILED DESCRIPTION:
The study will be conducted by the research team in close collaboration with the organization behind the multicomponent camps and their staff (Julemærkefonden/Julemærkehjem Hobro and Fjordmark). The multicomponent camps are well-established non-governmental institutions focusing on improving health and well-being in 7-14-year-old children by providing a structured environment, including social and physical activities, healthy meals and daily physical activities. Children of all weight classes can be referred to attend the camps by their general practitioner due to overweight, obesity and/or psychological challenges e.g., loneliness, bullying and family-related challenges. All 7-14-year-olds attend the camp free of charge.

In the present study, all participants will receive standard care during the 10-weeks at the multicomponent camp, which follows national recommendations concerning diet and physical activity. All participants will be screened for BED with the STOB screening tool before the intervention. Among those participants who screen positive for BED with the STOB screening tool, parents/guardians will be randomized to receive either:

Standard parental involvement during the camp (P-ST).

or

A parental BED intervention in addition to the standard parental involvement during the camp (P-BED)

In all cases where BED is suspected at recruitment based on the STOB screening tool, participants will be referred to a diagnostic interview (The Child Eating Disorder Examination (ChEDE)) to determine if participants fulfill the diagnostic criteria for BED. The use of ChEDE at baseline and after the intervention is implemented to validate the STOB screening-tool for future use. Therefore, a subsample of participants screened negative at recruitment with the STOB screening-tool (i.e., no BE behavior) will also undergo a diagnostic interview.

Throughout the study, interviews will be conducted with a subsample of participants, parents, and camp staff. Participants and camp staff will be interviewed to gain insights into their perspectives of using the STOB screening-tool. Moreover, parents will be interviewed to include their perspectives in the developmental process and to gain insights into their interpretation of the content, format, and perceived value of the parental BED intervention.

ELIGIBILITY:
Inclusion Criteria:

* Attending the camp in Hobro or Fjordmark from January 2027 to December 2027
* 7-14 years of age at recruitment
* Participants must have written informed consent from parent/guardian before camp to participate
* At least one parent/guardian submit written informed consent to participate in the study with their child

Exclusion Criteria:

* A medical condition affecting dietary intake and/or eating behavior
* Taking weight loss medication
* The parent/guardian don't understand the written informed consent
* Participant or parent/guardian are unwilling to or unable to comply with the study protocol and instructions given by the study staff.

Ages: 7 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 200 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2028-12 (Estimated); Study Completion 2036-01 (Estimated)

PRIMARY OUTCOMES:
Changes in Binge eating behavior using the STOB-screening tool | Baseline, 10-weeks (post-intervention), 10-12 weeks after the intervention, and 2 and 5 years after the intervention.
  The STOB-screening tool consist of five yes/no questions + one question about number of overeating episodes
Changes in prevalence of Binge eating disorder (BED) using the ChEDE | Baseline, and 10-weeks (post-intervention).
  Binge eating disorder will be assessed using the Child Eating Disorder Examination interview

SECONDARY OUTCOMES:
Changes in Body Mass Index standard deviation score (BMI-SDS) | Baseline, 10-weeks (post-intervention), 10-12 weeks after the intervention, and 2 and 5 years after the intervention.
  BMI-SDS calculated using World Health Organization Anthro-Plus software/cutoffs to define normal weight, overweight and obesity among participants.
Changes in Body fat (%) | Baseline, 10-weeks (post-intervention), and 2 and 5 years after the intervention.
  Measured in light clothing without shoes using a Bioelectric impedance (InBody model 270, Hopkins Medical Products, Grand Rapids, MI, USA).
Changes in Skeletal Muscle Mass (kg) | Baseline, 10-weeks (post-intervention), and 2 and 5 years after the intervention.
  Measured in light clothing without shoes using a Bioelectric impedance (InBody model 270, Hopkins Medical Products, Grand Rapids, MI, USA).

OTHER OUTCOMES:
Changes in Quality of Life using the PedsQL | Baseline, 10-weeks (post-intervention), 10-12 weeks after the intervention, and 2 and 5 years after the intervention.
  Quality of life (QoL) will be assessed using the Pediatric Quality of Life Inventory to assess total QoL, physical functioning, emotional functioning. social functioning, and school functioning.
Changes in appetitive traits using the CEBQ or AEBQ depending on age | Baseline, 10-weeks (post-intervention), 10-12 weeks after the intervention, and 2 and 5 years after the intervention.
  Appetitive traits will be measured using the Children's eating behavior questionnaire or Adult Eating behavior questionnaire depending on age to assess food responsiveness, emotional overeating/undereating, enjoyment of food, desire to drink, hunger, satiety responsiveness, slowness in eating, and food fussiness.

CONTACTS AND LOCATIONS:
Overall Officials: Jens M Bruun, Professor, Principal Investigator — University of Aarhus
Locations (2):
- Denmark (2):
  - Julemærkehjemmet Hobro, Hobro
  - Julemærkehjemmet Fjordmark, Kruså

IPD SHARING:
Plan to Share IPD: No